CLINICAL TRIAL: NCT05492747
Title: Does Kangaroo Care Have an Effect on Transition Time From Gavage Feeding to Full Oral Feeding in Premature Babies?
Brief Title: Kangaroo Care an EffectonTransitionTime From Gavage Feeding
Acronym: KangarooCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, DİDEM COŞKUN ŞİMŞEK, Principal Investigator, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Kangaroo Care on Oral Feeding
Record Dates: First submitted 2022-07-25; First posted 2022-08-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Premature Infants
Keywords: Gavage feeding; Kangaroo care; Oral feeding; Preterm babies
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kangaroo Care Effects on Feeding (Experimental): The researcher allocated the mothers blindly. Eligible mothers and their preterm babies were randomized to either the kangaroo care group or the standard care group (1:1) (Figure 1). The mothers' surnames were written and put in a bag. The surnames were drawn from the bag by lot. The lots were drawn by a neonatal nurse. Neonatal nurse is a research independent person. The first drawn surname was included in the kangaroo group, while the next one was included in the control group, respectively.
  Interventions: Other: Kangaroo Care an Effect

INTERVENTIONS:
Other: Kangaroo Care an Effect — Researchers evaluated vital signs and oxygen saturation of preterm infants in the kangaroo care group 15 minutes before kangaroo care. After the baby's mother was admitted to the NICU, she was assisted by the researcher for hand hygiene and they went to the incubator together. The mother was seated in a comfortable chair next to the incubator. After the researcher covered the head and back of the preterm baby with a baby blanket, she took it from the incubator and placed it between the mother's breasts, with the head up and upright. The baby was supported not only by the neck and shoulders, but also by the whole body. Skin contact between mother and baby was ensured at the highest level. The baby was positioned so that its lips were touching the mother's nipple. The researcher waited until the baby opened its mouth.

SUMMARY:
Objectives: Kangaroo care is a safe and effective alternative method to conventional neonatal care for newborn babies. The aim of this study was to evaluate the effect of kangaroo care on the transition time to full oral feeding in preterm infants fed by gavage.

Methods: This is a randomized controlled trial. This study was conducted in a level III neonatal intensive care unit of a university hospital in eastern Turkey 50 premature babies with a birth weight of ≥ 1000 g and a gestational age of 27-36 weeks, and their mothers were included in the study. The cases were randomly divided into two groups: kangaroo care, which would be applied up to five days a week, and standard care. Records of cases were kept regularly from their hospitalization until they reached full oral feeding.

DETAILED DESCRIPTION:
Study interventions i] Training: One day before starting the study, mothers in the kangaroo group were informed about kangaroo care. The training was provided in a meeting room outside the NICU. In the training, the advantages of the kangaroo care method for the mother and the baby and how the method will be applied were explained to the mothers. After the PowerPoint presentation, the mothers' questions were answered and they were given a kangaroo care guide prepared by the World Health Organization (WHO) [19].The training took about an hour. The researcher who provided the training is experienced in neonatal nursing and has a doctorate in pediatric nursing.

ii] Preparation of breast milk: The milks that the mothers milked and brought with storage bags were stored frozen below -18 degrees Celsius in the deep freezer of the food preparation room outside the NICU. These frozen milks were warmed by neonatal nurses according to the needs of the baby and given by syringe.

iii] Kangaroo care: Researchers observed vital signs and oxygen saturation of preterm infants in the kangaroo care group just before and during the kangaroo contact with the mother. After the baby's mother was admitted to the NICU, she was assisted by the researchers for hand hygiene and they went to the incubator together. The mother was seated in a comfortable chair next to the incubator. After the researchers covered the head and back of the preterm baby with a baby blanket, she took it from the incubator and placed it between the mother's breasts, with the head up and upright. The baby was supported not only by the neck and shoulders, but also by the whole body. Skin contact between mother and baby was ensured at the highest level. The baby was positioned so that its lips were touching the mother's nipple. The researchers waited until the baby opened its mouth. The baby's upper and lower lips were placed in such a way that the entire areola was in its mouth. The mother held her breast in a "C" shape with her hand. Thus, the baby's nose was prevented from being blocked. During the application, the researcher gave breast milk in the syringe to the baby through gavage. The babies and their mothers were observed by the researcher throughout the application. Kangaroo care was applied to the infants for 15-20 minutes during feeding, four times a day, five days a week. Kangaroo care of preterm infants fed by gavage continued until they achieved full oral feeding. Kangaroo care was also given to the babies who were connected to the ventilator.

iv] Standard care: Premature babies in this group were fed by gavage in the incubator. In standard neonatal care, parents could see their babies outside the incubator for 15-20 minutes. If parents want to touch their baby, they can do so through the open windows of the incubator, provided they wash their hands. Babies had only diapers and parents only touched their babies' hands, feet, back and abdomen without skin-to-skin contact. Ventilated premature babies are not placed on their parents' lap in accordance with NICU protocol.

v] Transition from gavage feeding to full oral feeding: The first feeding of preterm babies is usually made through the orogastric tube due to the incomplete development of sucking and swallowing reflexes and the immaturity of the gastrointestinal tract. Accordingly, premature babies included in the study were fed with an orogastric tube after a certain period of time after their hospitalization. Recordings were made daily and continued until the transition to full oral feeding was achieved.

ELIGIBILITY:
Inclusion Criteria:

* parents who agreed to participate in the study

Exclusion Criteria:

* healthy newborn
* congenital anomalies

Ages: 27 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
this study was measured the effects of kangaroo care in the transition period of preterm infants fed by gavage to full oral feeding. | 3 weeks
  Transition from gavage feeding to full oral feeding: The first feeding of preterm babies is usually made through the orogastric tube due to the incomplete development of sucking and swallowing reflexes and the immaturity of the gastrointestinal tract. Accordingly, premature babies included in the study were fed with an orogastric tube after a certain period of time after their hospitalization. Recordings were made daily and continued until the transition to full oral feeding was achieved.
  Questionnaire for switching to full oral feeding: It is a questionnaire in which the date of transition to full feeding of preterm infants is written.

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Coşkun Şimşek, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No